CLINICAL TRIAL: NCT05227729
Title: Descending Aorta Blood Flow to Guide Fluid Therapy During Surgery
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Torkjell Nostdahl, Principal investigator, Sykehuset Telemark
Other Study IDs: 264472
Record Dates: First submitted 2021-12-20; First posted 2022-02-07 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Hemodynamic Instability
Keywords: Hemodynamics; Blood Circulation; Aorta, Thoracic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing abdominal surgery: Inclusion criteria: > 18 years old, American Society of Anesthesiologists physical status 1-3, abdominal surgery of > 1,5 hrs estimated duration, no contraindications to the use of oesophageal ultrasound.
  Interventions: Diagnostic Test: Measurement of blood flow in descending aorta by suprasternal ultrasound Doppler technique; Diagnostic Test: Measurement of blood flow in descending aorta by transoesophageal ultrasound Doppler technique

INTERVENTIONS:
Diagnostic Test: Measurement of blood flow in descending aorta by suprasternal ultrasound Doppler technique — While study subjects are in general anesthesia the investigator will perform repeated measurements every 5 min.
Diagnostic Test: Measurement of blood flow in descending aorta by transoesophageal ultrasound Doppler technique — While study subjects are in general anesthesia the investigator will perform repeated measurements every 5 min.

SUMMARY:
The investigators will perform a clinical observational study of patients undergoing abdominal surgery. The study will be performed at Sykehuset Telemark, Skien. The aims of the study are to compare suprasternal and transoesophageal Doppler (reference method) to measure blood flow in the proximal descending aorta and to explore the variability of hemodynamic variables during surgery.

DETAILED DESCRIPTION:
Background and aim: The best validated method to estimate cardiac output with ultrasound requires measuring the Doppler velocity time integral (VTI) in the left ventricular outflow tract measured from the apical (lateral chest) window/ projection. However, this projection is often out of reach for anaesthesiologists during many surgical procedures (e.g. abdominal surgery) due to draping, and is often difficult to perform if the patient cannot be placed in the left lateral decubitus position. Alternatively, VTI in the proximal descending aorta may be measured via the suprasternal view, which is one of the standard projections in transthoracic echocardiography. This view is often available for anaesthesiologists during surgery on a patient in supine position. Assuming that changes in cardiac output are associated with changes in VTI in proximal descending aorta, this may provide the anaesthesiologist with a non-invasive measure of the response to a fluid challenge. The first aim of this study is to evaluate the ability of suprasternal Doppler to measure blood flow in the proximal descending aorta, and its agreement with the reference method oesophageal Doppler, during ongoing abdominal surgery.

Fluid challenges are typically given when stroke volume is reduced by 10-15%, which is considered a significant reduction. This is however dependent on the precision of the measurements, which is estimated during hemodynamic stability. During surgery, on the other hand, the variability may be larger, leading to erroneously concluding that stroke volume is reduced due to volume loss, when in fact this may be due to other stimuli related to surgery (mechanical, e.g. compression of large veins or the thoracic cavity, or stimuli affecting the autonomic nervous system, e.g. pain). The proportion of potentially falsely measured reduction may be calculated by performing repeated measurements during ongoing surgery. Thus, an other aim with this study is to explore the variability of measurements of stroke volume during surgery.

Study design: Clinical observational study.

Data collection: 30 patients scheduled to undergo laparoscopic or open abdominal surgical procedures (gastrointestinal or gynecological) of at least 1.5 hrs estimated duration. The patients should be of American Society of Anesthesiologists physical status 1-3 and have no contraindications to the use of oesophageal ultrasound. Hemodynamic data will be downloaded to a PC continuously from the clinical monitoring equipment (Philips Intellivue) using the VSCapture software (https://github.com/xeonfusion/VSCaptureMP) in VisualStudio (Microsoft). "Landmarks" in the procedure (e.g. surgical incision, manipulation in the surgical field and hemorrhage) will be recorded manually to relate the hemodynamic data to the different steps in the procedure. Blood flow velocity in the descending aorta will be measured using ultrasound machines in ordinary clinical use (GE Venue R 2.5; GE Healthcare). The Doppler recordings will be analyzed using commercially available software (EchoPAC; General Electric) after blinding.

Data analyzes:

* Considerations regarding sample size for agreement analyzes: The investigators will focus on within-subject variability, and the main outcome will be the corresponding within-subject limits of agreement. If both methods have a precision of 2.9%, limits of agreement will be 8.3%. Given 18 measurements per subject (one measurement every 5 min over 1.5 hrs), 25 subjects will give an 80% power for an upper confidence interval of the limits of agreement of 18%. By including 30 patients, the investigators allow for some unsuccessful measurements due to e.g. poor echogenicity.
* Considerations regarding sample size for variability analyzes: Given that the SD of oesophageal Doppler is 2.9%, the precision is 2.9%×1.96=5.7%. The probability of each evaluation of showing a false reduction is 0.8%. If surgery lasts 1.5 hrs with one evaluation every 5 min, the probability of at least one false reduction is 12%. If the precision is reduced with a doubled SD, the probability of at least one false reduction is 88%. Assuming a true SD of 2.9%; studying 25 subjects gives a power of 0.8 to detect a SD <3.0%.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo laparoscopic or open abdominal surgical procedures (gastrointestinal or gynecological) of at least 1.5 h estimated duration.
* The patients should be of American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* Pathology in the larynx, oesophagus or stomach
* Former surgery in larynx, oesophagus or stomach
* Thoracic aortic aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that plan to undergo abdominal surgery (gastrointestinal or gynecological) at Telemark hospital, Skien, Norway.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Change in blood flow velocity in descending aorta | During surgery, every 5 minutes. At least over a time period of 1,5 hours
  Suprasternal Doppler
Change in blood flow velocity in descending aorta | During surgery, every 5 minutes. At least over a time period of 1,5 hours
  Transoesophageal Doppler
Change in stroke volume | During surgery, every 5 minutes. At least over a time period of 1,5 hours
  Calculated from the measurements by transoesophageal Doppler

SECONDARY OUTCOMES:
Change in heart rate | During surgery, every 5 minutes. At least over a time period of 1,5 hours
  Measured in beats per minute, collected from standard monitoring device during surgery
Change in systemic vascular resistance | During surgery, every 5 minutes. At least over a time period of 1,5 hours
  Measured in dynes/second/cm^5. Calculated from the measurements by transoesophageal Doppler and standard monitoring device (mean arterial pressure)
Change in blood pressure | During surgery, every 5 minutes. At least over a time period of 1,5 hours
  Measured in mmHg, collected from standard monitoring device during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Torkjell Nøstdahl, MD, PhD, Principal Investigator — Telemark Hospital Trust
Locations (1):
- Telemark Hospital Trust, Skien, Vestfold Og Telemark, Norway